CLINICAL TRIAL: NCT04675801
Title: Safety and Efficacy of Bridging Antithrombotic Therapy During Elective Non-cardiac Surgery for Coronary Artery Disease Patients Treated With Oral Antiplatelet Agents
Brief Title: SAfety and EFficacy of Bridging Antithrombotic Therapy During Elective Non-cardiac Surgery
Acronym: SAFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, PhD, MD, Beijing Anzhen Hospital
Other Study IDs: SAFE
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
Keywords: Bridging antithrombotic therapy; Non-cardiac surgery; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bridging therapy with LMWH (n=475): Bridging therapy with LMWH was performed after discontinuation of oral antiplatelet agents prior to non-cardiac surgery
- Bridging therapy with tirofiban (n=475): Bridging therapy with tirofiban was performed after discontinuation of oral antiplatelet agents prior to non-cardiac surgery

SUMMARY:
Patients with coronary artery disease, especially after PCI, require long-term oral antiplatelet therapy. However, this patient population may inevitably require non-cardiac surgery for a variety of conditions. In order to avoid the occurrence of bleeding events, oral antiplatelet agents are usually discontinued before non-cardiac surgery in patients with coronary artery disease, which may increase the incidence of ischemic events. Therefore, it is important to provide patients with the optimal perioperative antithrombotic treatment to balance the risk of bleeding and ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Established coronary artery disease being treated with oral antiplatelet therapy
3. Non-cardiac surgery is planned and bridging antithrombotic therapy is considered necessary
4. Agree to participate in the study and provide written informed consent

Exclusion Criteria:

1. According to the consensus of Chinese experts on antiplatelet therapy in 2013, the surgical bleeding risk is low or extremely low
2. Requiring emergency non-cardiac surgery within 24 hours after admission
3. Currently being bleeding
4. Moderate or severe ischemic stroke or spontaneous intracranial hemorrhage in the past 6 months or traumatic intracranial hemorrhage in the past 1 year
5. Intracranial diseases or hemorrhagic diathesis
6. Contraindications for LMWH or GP IIb/IIIa receptor antagonists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Coronary artery disease patients treated with oral antiplatelet therapy are planned to undergo non-cardiac surgery with high or extremely high surgical bleeding risk
Sampling Method: Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | Perioperative period
  A composite of all-cause death, non-fatal myocardial infarction, or non-fatal stroke

SECONDARY OUTCOMES:
TIMI major or minor bleeding | Perioperative period
  A composite of major or minor bleeding events as defined by the TIMI bleeding criteria
Net adverse clinical events | Perioperative period
  A composite of major adverse cardiovascular events and TIMI major or minor bleeding
Net adverse clinical events | 30 days after surgery
  A composite of major adverse cardiovascular events and TIMI major or minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Liu, PhD, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No